CLINICAL TRIAL: NCT00387478
Title: A Double Blind Study to Investigate the Clinical Efficacy and Safety of TreeMATAMPL (Allergy Therapeutics, (UK) Ltd.), TreeMATA (Allergy Therapeutics, (UK) Ltd.) and Placebo in Patients With Seasonal Allergic Rhinitis Due to Birch Pollen Allergy, in an Environmental Exposure Chamber (EEC) Model When Exposed to Birch Pollen and Oak Pollen
Brief Title: Investigation of Efficacy and Safety of Tree MATAMPL,Tree MATA, and Placebo in Patients With Birch-Induced Seasonal Allergic Rhinitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollement target could not be achieved, study will not resume
Sponsor: Allergy Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TreeMATAMPL204; P2DP06002
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Type I Hypersensitivity
Keywords: Allergy; Specific Immunotherapy; Tree; Environmental Exposure Chamber
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): modified Tree pollen allergen absorbed to Tyrosine and containing MPL adjuvant
  Interventions: Biological: Tree MATA MPL or Tree MATA
- 2 (Experimental): modified Tree pollen allergen absorbed to Tyrosine
  Interventions: Biological: Tree MATA MPL or Tree MATA
- Placebo (Placebo Comparator): 4 injections of placebo 0.5 ml (2% tyrosine)
  Interventions: Biological: Tree MATA MPL or Tree MATA

INTERVENTIONS:
Biological: Tree MATA MPL or Tree MATA — 4 injections of increasing dose strength for Tree MATA MPL or Tree MATA:
  1. 600 SU/0.5 ml
  2. 1600 SU/0.5 ml
  3. 4000 SU/0.5 ml
  4. 4000 SU/0.6 ml
  4 injections of 0.5 mL of 2% w/v L-tyrosine for Placebo

SUMMARY:
Tree MATAMPL has been developed to provide pre-seasonal specific immunotherapy for patients with hypersensitivity to Tree (birch, alder, hazel) pollen (hay fever). This novel formulation is designed to provide a vaccine that will be efficacious with only four escalating dose injections administered before the start of the pollen season. In this Study the Efficacy will be assessed by exposing allergic subjects to birch pollen in an environmental exposure chamber EEC. Patient symptomatic response to birch pollen and patient quality of life in the EEC will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be male or female and aged 18 to 50 years inclusive.
* Patients must have at least a two-year clinical history of SAR due to birch pollen allergy.
* Patients must have allergy to tree pollen allergen, defined by positive case history and positive skin prick test for tree pollen allergen (wheals of ≥ 5 mm (birch) and ≥ 3 mm (hazel and alder) greater than the negative control after skin prick testing) at Visit 1. Patients who will be skin tested at Visit 1 must adhere to the washout time for antihistamines.
* Specific IgE for birch tree pollen as documented by a radioallergosorbent test (RAST), or equivalent test, with class ≥ 2.
* Patients must obtain minimum qualifying symptom scores on the final two pre-treatment birch pollen exposure sessions (Visits 4 and 5) to be enrolled into the study. Minimum qualifying symptom scores are defined as a TSS of at least 12 out of a possible 24 and a NSS of at least 7 out of a possible 12 on at least one symptom diary card on each of Visits 4 and 5. Furthermore, a minimum priming criteria for NSS of 7 out of a possible 12, including a score of at least 2 for runny nose, on two diary cards during each of Visits 4 and 5, must be obtained.
* Patients must observe the drug washout times prior to Screening (Visit 1). The use of other medications will be permitted if they are not expected to interfere with the ability of the patient to participate in the study and provided they have been on a stable regimen (i.e., the same dosage and administration) for six weeks prior to Screening.
* Males or non-pregnant, non-lactating females who are post-menopausal or naturally or surgically sterile (hysterectomy; bilateral oophorectomy; bilateral tubal ligation with surgery at least 6 weeks prior to study initiation). Postmenopausal is defined as at least 12 months natural spontaneous amenorrhea, or at least six weeks following surgical menopause (bilateral oophorectomy). Females of childbearing potential should be using one of the following acceptable birth control methods:Intrauterine device (IUD) in place for at least 3 months;Barrier method (condom or diaphragm) with spermicide; Stable hormonal contraceptive for at least 3 months prior to study and through study completion;Abstinence; Non-heterosexual lifestyle.
* Patients who are normally active and otherwise judged to be in good health on the basis of medical history, physical examination and routine laboratory tests.
* Patients must be willing and able to give written informed consent and must provide this consent.
* Patients must be willing and able to attend required study visits. 11.Patients must be able to follow instructions.

Exclusion Criteria:

A patient will not be included in this study if one or more of the following criteria apply:

* Have a positive skin prick test [wheal (longest diameter) ≥ 3 mm greater than the negative control] at Visit 1 to any of the following perennial allergens: house dust mites (Dermatophagoides pteronyssinus and Dermatophagoides farinae), molds (Cladosporium cladosporioides, Alternaria alternata, Penicillium chyrsogenum (notatum), and Aspergillus fumigatus), or epithelia (cat, dog, and horse). In these cases, a careful history is to be taken and if moderate or severe symptoms are reported when exposed to the aforementioned allergens, the subject is to be excluded. Exception: the source of the allergen (cat, dog, horse) can be avoided for the entire study. Subjects with mild or no symptoms when exposed to the aforementioned allergens during the 3 years prior to Visit 1 will be allowed to enroll. Mild symptoms are defined as: sign/symptom clearly present, but minimal awareness, easily tolerated.
* Concurrent disease that might complicate or interfere with investigation or evaluation of the study medications or the skin prick test result, such as:

Rhinitis medicamentosa; Large obstructive nasal polyps; Documented evidence of acute or significant chronic sinusitis, or upper respiratory tract infection as determined by the individual Investigator; Asthma, with the exception of mild intermittent asthma, to lessen confounding by asthma medications; History of hospitalization for asthma; History or presence of acute or subacute atopic dermatitis, chronic dermatitis, urticaria factitia, or urticaria due to physical/chemical influence.

* Current diagnosis of seasonal asthma caused by tree pollen exposure.
* Concurrent use or inadequate washout of any prohibited medication.
* Chronic or intermittent use of inhaled, nasal, ocular, oral, intramuscular, intravenous, or potent or super-potent topical corticosteroids (as assessed by the Investigator).
* Chronic use of long acting antihistamines and other concomitant medications (e.g., tricyclic antidepressants) that would affect assessment of the effectiveness of study drug(s).
* Are pregnant or lactating.
* Any systemic disorder that could interfere with the evaluation of the study medication(s).
* Upper or lower respiratory infection requiring antibiotics within 14 days of Visit 2.
* Diagnosis of sinusitis within 30 days of Visit 2.
* Any ocular disorder (other than allergic conjunctivitis) including presumed infectious ocular disease (bacterial, fungal, viral, etc.), which could interfere with the evaluation of the study medication.
* Hypersensitivity to the study drug(s) excipients.
* Patients with active or quiescent tuberculous infection of the respiratory tract, untreated local or systemic fungal or bacterial or systemic viral infections or parasitic or ocular herpes simplex.
* Patients who have experienced nasal septal ulcers, nasal surgery or nasal trauma within 90 days of enrollment into this study.
* Clinical history of anaphylaxis or idiopathic anaphylaxis.
* Patients with a clinical history of immunodeficiency, including those who are on immunosuppressant therapy.
* Patients with an auto-immune disease (e.g. of liver, kidney, thyroid, nervous system)
* Patients with a history of angioedema
* Patients in whom tyrosine metabolism is disturbed, especially in the case of tyrosinemia and alkaptonuria.
* Patients with contraindications to adrenaline.
* Patients taking β-blockers, including eye drops, for any indication.
* Patients taking Monoamine Oxidase Inhibitors
* Current diagnosis of chickenpox or measles.
* Clinical history of drug or alcohol abuse which would, at the Investigator's discretion, interfere with the patient's participation in the study.
* Clinical history of severe or uncontrolled cardiovascular, pulmonary, hepatic, renal and/or other disease/illness that could be expected to interfere with the study.
* Clinical history, or evidence, of nasolacrimal drainage system malfunction.
* Study site staff or immediate relatives of study site staff or other individuals who would have access to the clinical study protocol.
* Patient that has received TreeMATAMPL in any previous clinical trial.
* History of immunotherapy with tree pollen extract, except if treatment was successfully completed 3 years prior to Visit 1 and SAR symptoms had reappeared prior to Visit 1.
* Patient received treatment with preparation containing MPL during the past 12 months.
* Participation in any other investigational study within 30 days before Visit 1 or concomitantly with this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Assess the clinical efficacy as measured by Total Symptom Scores (TSS) of TreeMATAMPL versus placebo in reducing Allergic Rhinitis (AR) symptoms caused by birch tree pollen in an Environmental Exposure Chamber (EEC) Model. | about 10 weeks

SECONDARY OUTCOMES:
Assess the clinical efficacy of TreeMATAMPL versus placebo and TreeMATA in reducing AR symptoms caused by birch and oak tree pollen in an EEC model | about 10 weeks
Assess the responder/non-responder rate in TSS, NSS and NNSS of TreeMATAMPL versus placebo and TreeMATAMPL versus TreeMATA | about 10 weeks
Evaluate the correlation between TSS obtained during the baseline birch EEC session compared to baseline oak EEC session | about 10 weeks
Evaluate the correlation between the TSS change observed (baseline to post treatment) during the birch EEC sessions compared to oak EEC sessions | about 10 weeks
Assess the correlation between the percentage of positive skin prick test results between birch pollen and the following tree pollen: Oak, ash, red maple, poplar, black walnut, beech, sycamore and American elm | during screening period (normally 1 day)
Assess the immunological response to TreeMATAMPL versus placebo and for TreeMATAMPL versus TreeMATA immunotherapy in patients with SAR. | IgG (IgG/IgG4) levels will be assessed after V1, 14, 21
Evaluate the impact of TreeMATAMPL versus placebo and for TreeMATAMPL versus TreeMATA on quality-of-life in patients with SAR using the Rhinoconjunctivitis Quality of Life Questionnaire for use in the EEC. | about 10 weeks
Assess the safety and tolerability of TreeMATAMPL versus placebo and TreeMATAMPL versus TreeMATA in patients with SAR. | about 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, CCFP, Principal Investigator — Allied Research International Inc, Mississauga, Canada
Locations (1):
- Allied Research International Inc., Mississauga, Ontario, Canada